CLINICAL TRIAL: NCT04078581
Title: Profiling Fecal Samples to Optimize Selection of Stool Donors for Fecal Microbiota Transplantation
Brief Title: Profiling Fecal Samples for Selection of Donors of Feces
Acronym: PROFIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP190341; 2019-A01012-55 (Other: ANSM)
Record Dates: First submitted 2019-04-26; First posted 2019-09-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2020-03

CONDITIONS: Fecal Microbiota Transplantation
Keywords: Selection of healthy donors; Healthy volunteers; Stool donors; Fecal microbiota transplantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy controls (Experimental): Questionnaire and fecal sample collection
  Interventions: Other: Questionnaire and fecal sample collection

INTERVENTIONS:
Other: Questionnaire and fecal sample collection — Questionnaire and fecal sample collection in order to select donors for FMT.

SUMMARY:
Fecal microbiota transplantation (FMT) represents a promising therapeutic in numerous clinical situations associated with dysbiosis. Today, this procedure is recommended in patients with recurrent Clostridioides difficile infections but beneficial effects of FMT have also been described in other diseases associated with intestinal dysbiosis …. A donor effect which could be related to the inter-individual variability of microbiota and microbiome leading to specific metabolic capacities may influence the efficacy of the procedure.

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) represents a promising therapeutic in numerous clinical situations associated with dysbiosis. Today, this procedure is recommended in patients with recurrent Clostridioides difficile infections but beneficial effects of FMT have also been described in other diseases associated with intestinal dysbiosis …. A donor effect which could be related to the inter-individual variability of microbiota and microbiome leading to specific metabolic capacities may influence the efficacy of the procedure. The aim of our study is to measure fecal biochemical, microbial and immunological parameters that are known to influence gut homeostasis in a group of 40 healthy donors to establish a referential profile of human stools to optimize donor profiling, beyond the infectious parameters, to increase the success rate of FMT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Healthy volunteers
3. Participant having been informed of the study and having sign a consent to participation
4. Patient affiliated with a social security or beneficiary of such a social protection

Exclusion Criteria:

1. Person subject to legal protection (guardianship, trusteeship, etc.)
2. Chronic disease that can alter the intestinal microbiota: cancer or malignant disease, bowel disease, diabetes, hypertension, hypercholesterolemia, ....
3. Presence in the 1st degree family of one of the chronic diseases mentioned above
4. Blood in stools
5. Chronic drug treatment likely to alter the intestinal microbiota
6. Travel to a tropical country in the last 3 months or extended stay (> 3 months) for less than 1 year
7. Hospitalization abroad (> 24h) in the last 12 months
8. Hospitalization abroad (> 24h) of a family member living under the same roof during the last 12 months
9. Medical consultation in the last 3 months (other than administrative)
10. Contact with a person with an infectious or contagious disease for more than 3 months
11. Digestive disorders / febrile gastroenteritis (diarrhea with fever) in the last 3 months
12. Febrile illnesses for more than 3 months
13. Antibiotic treatment in the last 3 months
14. Treatment with PPIs in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Dosage of fecal samples with search for differentiated fecal profiles. | At 12 months
  16S genomic analysis of microbiota will be performed for the evaluation of alpha and beta diversities of microbiota.
  Results will be aggregated to define differentiated faecal profiles in healthy volunteers.

SECONDARY OUTCOMES:
Dosage of fecal biomarkers with search for differentiated fecal profiles. | At 12 months
  Fecal biomarkers such as calprotectin will be dosed. Results will be aggregated to define differentiated faecal profiles in healthy volunteers.
Quantification of colonic inflammation in mouse model. | At 15 months
  The quantification of colonic inflammation by myeloperoxidase assay using a sandwich ELISA enzyme-linked immunosorbent assay.
  Mouse model : authorization APAFlS#7600-20l60620l6336853 v3

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KAPEL, PharmD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No